CLINICAL TRIAL: NCT01167309
Title: LEO 27847 - Safety, Tolerability, Pharmacokinetic and Pharmacodynamic Study in Secondary Hyperparathyroidism Patients With Chronic Kidney Disease
Brief Title: LEO 27847 - Safety, Tolerability, Pharmacokinetic and Pharmacodynamic Study in Secondary Hyperparathyroidism Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: LEO Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Other
Other Study IDs: LEO 27847-S02
Record Dates: First submitted 2010-07-02; First posted 2010-07-22 (Estimated); Last update posted 2025-02-24 (Actual); Status verified 2013-10

CONDITIONS: Secondary Hyperparathyroidism
Keywords: Safety and tolerability of LEO 27847
MeSH Terms: conditions — Hyperparathyroidism, Secondary

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (5):
- Part 1 SAD (Active Comparator): four diffferent doses
  Interventions: Drug: LEO 27847
- Part 2a MAD (Placebo Comparator): three doses
  Interventions: Drug: LEO 27847
- Part 2b (Active Comparator): 0.24 mg LEO 27847
  Interventions: Drug: LEO 27847
- Part 2c (Active Comparator): 0.24 mg LEO 27847
  Interventions: Drug: LEO 27847
- Parat 2a MAD (Placebo Comparator): one dose
  Interventions: Drug: LEO 27847

INTERVENTIONS:
Drug: LEO 27847 — First in patient

SUMMARY:
The purpose of this trial is to determine the safety and tolerability of ascending single and multiple oral doses of LEO 27847 in secondary hyperparathyroidism patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 to 75 years (inclusive) at screening.
* Patients with body mass index within 18 to 34 kg/m2 (inclusive).
* Haemoglobin is stable (≥9 g/dL or 5.6 mmol/L)
* Parathyroid hormone (PTH) is ≥200 pg/mL and <800 pg/mL.
* Screening serum albumin is ≥30 g/L.
* C-reactive protein <25 mg/L.

Exclusion Criteria:

* Adjustment of vitamin D sterols within 14 days before the screening visit and patients for whom adjustment of vitamin D sterols is planned from screening until end of study.
* Adjustment of calcium supplements within 14 days before the screening visit and patients for whom adjustment of calcium supplements is planned from screening until end of study.
* Adjustment of phosphate binder within 14 days before the screening visit and patients or whom adjustment of phosphate binder is planned from screening until end of study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2010-06; Primary Completion 2011-10 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Safety and Tolerability | 7 days after last dosing
  Adverse events, vital signs, ECG, laboratory evaluation, physical examination

SECONDARY OUTCOMES:
Pharmacokinetics and Pharmacodynamics | 7 days after last dosing
  LEO 27847, PTH, calcium, Vitamin D and phosphate in blood. LEO 27847 in urine

CONTACTS AND LOCATIONS:
Overall Officials: Medical Expert, Study Director — LEO Pharma
Locations (2):
- CRS Clinical Research Services Kiel GmbH, Kiel, Germany
- Centralny Szpital Kliniczny MON, Warsaw, Poland

IPD SHARING:
Plan to Share IPD: No